CLINICAL TRIAL: NCT05125211
Title: A PhaseⅠRandomised, Double-blind, Placebo-controlled, Study to Evaluate the Safety, Tolerability, and Pharmacokinetics Characteristics of the Oral Topical Use of GB001 Recombinant Peptide Spray in Chinese Healthy Adult Subjects
Brief Title: Safety,Tolerability,and Pharmacokinetics Profiles of GB001 Recombinant Peptide Spray in Healthy Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Echon Biopharm Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YK2019L01P-Ⅰ
Record Dates: First submitted 2021-10-24; First posted 2021-11-18 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single dose-escalation of GB001 recombinant peptide spray (Experimental): Each subject will receive one single administration of GB001 recombinant peptide. The dosage of each group is 0.054mg, 0.108mg, 0.216mg, 0.432mg and 0.864mg, respectively.
  Interventions: Drug: GB001 recombinant peptide spray; Drug: Placebo
- Oral retention time test for a single dose (Experimental): Each subject will receive one single administration of GB001 recombinant peptide. The dosage of the group is 0.108mg.
  Interventions: Drug: GB001 recombinant peptide spray
- Multiple Ascending Dose of GB001 recombinant peptide spray (Experimental): Each subject will be dosed with oral spray of GB001 recombinant peptide ten times per day for four days. GB001 recombinant peptide will be administrated, and the dosage of each group is 0.108mg, 0.216mg and 0.432mg, respectively.
  Interventions: Drug: GB001 recombinant peptide spray; Drug: Placebo

INTERVENTIONS:
Drug: GB001 recombinant peptide spray — administrated oral spray
Drug: Placebo — administrated oral spray
  Arms: Multiple Ascending Dose of GB001 recombinant peptide spray; Single dose-escalation of GB001 recombinant peptide spray

SUMMARY:
This trial is conducted in China. The aim of this clinical trial is to assess the safety , tolerability and pharmacokinetics profiles of GB001 by single ascending dose and multiple ascending doses in healthy subjects after topical buccal delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females aged 18 to 45 years, with a body mass index(BMI) 19-26kg/m2 and body weight no less than 45 kg (female) or 50 kg (male).
2. The results in the screening examinations (including general physical examination, vital signs, laboratory examinations, electrocardiogram, chest radiograph, etc.) are in the normal range, or are abnormal without clinical significance assessed by the investigator.
3. Subjects and their sexual partners agree to take effective contraceptive measures during the study period and at least 3 days after the end of the study.
4. Understanding and willing to comply strictly with the clinical trial protocol, complete all test procedures required in this trial, understand and sign informed consent form.

Exclusion Criteria:

1. Those allergic to GB001 peptide or any other drugs, or suffered from allergic disease or allergic constitution.
2. Any obvious clinical symptoms or abnormal test results with clinical significance suggested organ or system illness, unsuitable for inclusion in this trial in the investigator's judgement.
3. Subjects has obvious oral lesions or diseases, such as erosion of oral mucosa, ulcer or obvious periodontitis.
4. The weekly alcohol intake in 90 days before screening is more than 21 units (male) and more than 14 units (female) , or the subject is unwilling to stop drinking whenever required for the trial procedure.
5. Subject who smoke more than 10 cigarettes per day or is unwilling to stop smoking whenever required for the trial procedure.
6. Subject with a history of drug abuse, or those with positive urine screening test for drug abuse.
7. Subject who use of any other drugs within 30 days prior to screening, including prescription drugs, non-prescription drugs, biologicals, vitamins, minerals and nutritional supplements.
8. Blood loss or blood donation more than 400 mL within 90 days prior to screening.
9. Received major surgery within 90 days prior to screening, or participated in any other drug/device clinical trial.
10. Pregnant or lactating women; or female subject of childbearing age have a positive serum pregnancy test result during the screening.
11. Subject with dizzy needle or difficulty in venous blood collection.
12. Subject unsuitable for the trial in the judgement of the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Through the study completion, an average of 2 weeks
  The number and the incidence of serious and non-serious adverse events observed in each treatment will be used to assess the safety and tolerability

SECONDARY OUTCOMES:
Pharmacokinetics Characteristics， t½ of GB001 recombinant peptide | Up to 240 minutes after last dose
  Apparent terminal phase half-life
Pharmacokinetics Characteristics , Cmax of GB001 recombinant peptide | Up to 240 minutes after last dose
  Maximum plasma concentration
Pharmacokinetics Characteristics , Tmax of GB001 recombinant peptide | Up to 240 minutes after last dose
  Time of maximum plasma concentration
Pharmacokinetics Characteristics , AUC of GB001 recombinant peptide | Up to 240 minutes after last dose
  Area under the plasma concentration versus time curve
Pharmacokinetics Characteristics , Vd of GB001 recombinant peptide | Up to 240 minutes after last dose
  Apparent distribution volume
Pharmacokinetics Characteristics , Ctrough of GB001 recombinant peptide | Up to 240 minutes after last dose
  Trough plasma concentration

OTHER OUTCOMES:
Oral retention time | Up to 120 minute after first dose
  Oral retention time

CONTACTS AND LOCATIONS:
Overall Officials: Feng Shao, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No